CLINICAL TRIAL: NCT00571935
Title: Efficacy and Safety of Insulin Aspart in MDI or CSII in Children Below 7 Years of Age With Type 1 Diabetes Mellitus
Brief Title: Efficacy and Safety of Insulin Aspart in MDI or CSII in Children Below 7 Years of Age With Type 1 Diabetes
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ANA-1507
Record Dates: First submitted 2007-12-11; First posted 2007-12-12 (Estimated); Last update posted 2016-12-21 (Estimated); Status verified 2016-12

CONDITIONS: Diabetes; Diabetes Mellitus, Type 1
MeSH Terms: conditions — Diabetes Mellitus; Diabetes Mellitus, Type 1 | interventions — Insulin Aspart

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: insulin aspart
Drug: soluble human insulin

SUMMARY:
This trial is conducted in Europe.

The aim of this trial is to investigate the efficacy of insulin aspart compared to soluble human insulin on blood glucose control in children below 7 years of age with type 1 diabetes.

ELIGIBILITY:
Inclusion Criteria:

* Type 1 diabetes for at least 1 year
* HbA1c below 12.0%
* Treatment with regular human insulin and insulin NPH for at least 1 month
* Receive more than 2 injections daily

Exclusion Criteria:

* Receipt of investigational product within 6 months prior to trial participation
* Known or suspected allergy to investigational product
* Receipt of of insulin aspart within 3 months prior to trial participation

Max Age: 7 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 61 (Actual)
Dates: Start 2003-08; Primary Completion 2004-10 (Actual); Study Completion 2004-10 (Actual)

PRIMARY OUTCOMES:
HbA1c | after 26 weeks of treatment

SECONDARY OUTCOMES:
Overall glycaemic control
Occurrence of adverse events
Occurrence of serious adverse events
Frequency of hypoglycaemia episodes
Quality of Life (QoL)

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Registry (GCR, 1452), Study Director — Novo Nordisk A/S
Locations (5):
- Poland (5):
  - Novo Nordisk Investigational Site, Bialystok
  - Novo Nordisk Investigational Site, Gliwice
  - Novo Nordisk Investigational Site, Kielce
  - Novo Nordisk Investigational Site, Krakow
  - Novo Nordisk Investigational Site, Warsaw

REFERENCES:
- [Result] Pankowska E, Nazim J, Szalecki M, Urban M. Equal metabolic control but superior caregiver treatment satisfaction with insulin aspart in preschool children. Diabetes Technol Ther. 2010 May;12(5):413-8. doi: 10.1089/dia.2009.0155. PMID 20388052
- See also: Clinical Trials at Novo Nordisk — http://novonordisk-trials.com